CLINICAL TRIAL: NCT00847080
Title: Treatment With Sitagliptin Phosphate in Patients With Reactive Hypoglycemia Secondary to Dysinsulinism. A Controlled, Randomized, Double-blind, Clinical Trial
Brief Title: Treatment With Sitagliptin for Reactive Hypoglycemia Secondary to Dysinsulinism
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Francisco J Gomez-Perez, Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MK-0431
Record Dates: First submitted 2009-02-18; First posted 2009-02-19 (Estimated); Last update posted 2011-04-26 (Estimated); Status verified 2009-02

CONDITIONS: Reactive Hypoglycemia
Keywords: Reactive hypoglycemia; Sitagliptin; Glucagon-Like Peptide 1; Incretins; Prediabetes
MeSH Terms: conditions — Hypoglycemia; Prediabetic State | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sitagliptin (Experimental)
  Interventions: Drug: Sitagliptin phosphate
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sitagliptin phosphate — Sitagliptin phosphate 100 mg per day per 2 weeks
  Other Names: Januvia
  Arms: Sitagliptin
Drug: Placebo — Placebo 1 tablet per day per 2 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether sitagliptin is effective in the treatment of reactive hypoglycemia by dysinsulinism.

DETAILED DESCRIPTION:
Symptomatic reactive hypoglycemia is an abnormal glucose decrease after meal ingestion. Patients with this abnormality as an early manifestation of glucose intolerance are at higher risk of type 2 diabetes. The pathophysiology of this abnormality appears to be related with delayed first phase insulin release. Improvement of first phase insulin secretion and delay in gastric emptying induced by sitagliptin phosphate could have favorable effects in patients in whom delayed insulin secretion is associated with reactive hypoglycemia.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and biochemical diagnosis of prediabetic reactive hypoglycemia
* Must be able to swallow tablet
* Negative pregnancy test (when appropriate)

Exclusion Criteria:

* Renal insufficiency
* Hepatic insufficiency
* Diabetes (any type)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2008-12; Primary Completion 2010-12 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Clinical improvement assessed by a validated questionnaire | 2 weeks

SECONDARY OUTCOMES:
Glucose, insulin, GLP1, GIP | First and last evaluations

CONTACTS AND LOCATIONS:
Overall Officials: Francisco J Gomez-Perez, MD, Principal Investigator — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Locations (1):
- Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran, Mexico City, Mexico City, Mexico

REFERENCES:
- See also: Click here for information of the study location — http://www.innsz.mx/opencms/contenido/english.html
- See also: Click here for information of study sponsor in english — http://www.merck.com/